CLINICAL TRIAL: NCT01298934
Title: A Phase I/II Open Label Study of LBH589, a Novel Histone Deacetylase Inhibitor (HDACi), in Patients With Primary Myelofibrosis (PMF) and Post-polycythemia/Essential Thrombocythemia Myelofibrosis (Post-PV/ET MF)
Brief Title: LBH589 (Panobinostat) for the Treatment of Myelofibrosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ronald Hoffman (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Ronald Hoffman, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 08-0572; LBH589-JM
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Primary Myelofibrosis; Polycythemia Vera, Post-Polycythemic Myelofibrosis Phase; Post-Essential Thrombocythemia Related Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis; Polycythemia Vera | interventions — Panobinostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LBH589 (Experimental): Dose escalation study starting at 20mg by mouth three times a week, given weekly for 24 weeks in the phase I portion of the study.
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — Dose escalation study starting at 20mg by mouth three times a week, given weekly for 24 weeks in the phase I portion of the study.
  Other Names: Panobinostat

SUMMARY:
LBH589 is an oral drug that targets the myelofibrosis cells in the bone marrow and induces cell death by allowing for the expression of certain suppressed genes that are important in regulating cell survival. Based on laboratory studies, the hypothesis is that this drug will selectively kill the stem cells responsible for causing myelofibrosis and result in reduction in spleen size and ultimately restoration of normal bone marrow function.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥ 18 years old
2. Ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
3. Newly diagnosed MF with intermediate or high risk Lille Scoring System (Hb<10g/dL, WBC <4.0 or >30 X 109/L; risk group 1=intermediate and 2= high), or symptomatic splenomegaly that is >10cm below costal margin.
4. Previously treated MF that are refractory, intolerant or relapsed in disease
5. Patients must meet the following laboratory criteria:

   * ANC ≥ 1.0 x 109/L
   * Platelets ≥ 60 x 109/L
   * Calculated CrCl ≥ 45 mL/min (MDRD Formula)
   * AST and ALT ≤ 2.5 x ULN
   * Serum bilirubin < 1.5 x ULN
   * Albumin > 3.0 g/dl
   * Serum potassium ≥ LLN
   * Total serum calcium [corrected for serum albumin] or ionized calcium ≥LLN,
   * Serum magnesium ≥ LLN
   * Serum phosphorus ≥ LLN
   * TSH ≤ ULN and free T4 within normal limits. Patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism.
6. Baseline MUGA or ECHO must demonstrate LVEF ≥ the lower limit of the institutional normal.
7. ECOG Performance Status of ≤ 2

Exclusion Criteria:

1. Prior HDAC, DAC, HSP90 inhibitors or valproic acid for the treatment of cancer
2. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to first LBH589 treatment
3. Peripheral neuropathy > 1
4. Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

   * Patients with congenital long QT syndrome
   * History or presence of sustained ventricular tachyarrhythmia.(Patients with a history of atrial arrhythmia are eligible but should be discussed with the Sponsor prior to enrollment)
   * Any history of ventricular fibrillation or torsade de pointes
   * Bradycardia defined as HR< 50 bpm. Patients with pacemakers are eligible if HR ≥ 50 bpm.
   * Screening ECG with a QTc > 450 msec
   * Right bundle branch block + left anterior hemiblock (bifascicular block)
5. Patients with myocardial infarction or unstable angina ≤ 6 months prior to starting study drug
6. Other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV , uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
7. Impairment of GI function or GI disease that may significantly alter the absorption of LBH589
8. Patients with diarrhea > CTCAE grade 1
9. Other concurrent severe and/or uncontrolled medical conditions (e.g., uncontrolled diabetes or active or uncontrolled infection) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol
10. Patients using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
11. Concomitant use of CYP3A4 inhibitors
12. Patients who have received targeted agents within 2 weeks or within 5 half-lives of the agent and active metabolites (which ever is longer) and who have not recovered from side effects of those therapies.
13. Patients who have received chemotherapy within 3 weeks; or radiation therapy to > 30% of marrow-bearing bone within 3 weeks prior to starting study treatment; or who have not yet recovered from side effects of such therapies.
14. Patients with an active bleeding tendency or are receiving any treatment with therapeutic doses of sodium warfarin (Coumadin®) or coumadin derivatives. Low doses of Coumadin® (e.g. ≤ 2 mg/day) to maintain line patency (if applicable) is allowed.
15. Patients who have undergone major surgery ≤ 4 weeks prior to starting study drug or who have not recovered from side effects of such therapy
16. Women who are pregnant or breast-feeding or women of childbearing potential (WOCBP) not using an effective method of birth control. WOCBP are defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months). Women of childbearing potential must have a negative serum pregnancy test within 24hrs of receiving the first dose of study medication.
17. Male patients whose sexual partners are WOCBP not using effective birth control
18. Patients with a prior malignancy with in the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix)
19. Patients with known positivity for human immunodeficiency virus (HIV) ) or hepatitis C; baseline testing for HIV and hepatitis C is not required
20. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff.
21. Disease associated with secondary MF such as metastatic carcinoma, lymphoma, myelodysplasia, hairy cell leukemia, mast cell disease or acute leukemia (including M7 disease or acute panmyelosis with MF)
22. Presence of chromosomal translocation t(9:22) or molecular BCR/ABL rearrangement as detected by RT-PCR in bone marrow or peripheral blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of oral LBH589 in patients with PMF, post-PV/ET MF | 28 days
  Phase I
Evaluation of treatment response by International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) | 6 months
  Phase II

SECONDARY OUTCOMES:
Assess changes in biomarkers | 6 months
  JAK2V617F allele burden H3/H4 acetylation status peripheral blood CD34+ stem cell burden CXCR4 expression on CD34+ peripheral blood stem cells

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Hoffman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States